CLINICAL TRIAL: NCT07153042
Title: National Implementation of an Evidence-Based HIV Prevention Program: Multilevel Scale-Up Strategies and Precision Prevention
Brief Title: Sustainability and Precision Prevention Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Ministry of Health, Bahamas (Unknown)
Responsible Party: Principal Investigator, Bo Wang, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002463
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Sustainability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1 (Experimental): All grade six teachers will go through the Usual Implementation (UI) of FOYC+CImPACT (teacher training only in Year 1).
  Interventions: Behavioral: FOYC+CImPACT
- Stage 2 (Experimental): Based on their performance in Year 1, teachers who do not meet the benchmark (implementing > 80% of core activities) will be randomized to receive 1) "Biweekly Monitoring and Feedback (BMF)" or 2) "BMF+Site-Based Assistance Mentorship (SAM)." Responders (completing at least 80% of core activities) will continue with UI.
  Interventions: Behavioral: Biweekly monitoring and feedback (BMF); Behavioral: Site-based assistance and mentorship (SAM); Behavioral: FOYC+CImPACT
- Stage 3 (Experimental): At the end of Year 2 (stage 2), the performance of the teachers in all three intervention arms will be assessed again. Non-responders in the UI arm will be re-randomized to receive either BMF or BMF+SAM. Non-responders in the BMF-only group will be re-randomized to receive BMF+SAM or BMF+enhanced SAM. Non-responders in the BMF+SAM group will receive BMF+enhanced SAM.
  Interventions: Behavioral: Biweekly monitoring and feedback (BMF); Behavioral: Site-based assistance and mentorship (SAM); Behavioral: Enhanced site-based assistance and mentorship (Enhanced SAM); Behavioral: FOYC+CImPACT

INTERVENTIONS:
Behavioral: Biweekly monitoring and feedback (BMF) — School coordinators will monitor teachers' implementation progress biweekly and provide feedback to teachers.
  Arms: Stage 2; Stage 3
Behavioral: Site-based assistance and mentorship (SAM) — High-performing teachers will serve as team leaders and guide non-responding teachers on preparation and planning. The team leader will promote group activities and enhance interaction among teachers in these meetings.
  Arms: Stage 2; Stage 3
Behavioral: Enhanced site-based assistance and mentorship (Enhanced SAM) — A FOYC coach (with FOYC implementation and training experience) will provide tailored in-person support, facilitate goal-setting, opportunities to interact with consultants, supportive text messaging, continuing education, networking strategies, and monthly check-ins.
  Arms: Stage 3
Behavioral: FOYC+CImPACT — Focus on Youth in the Caribbean (FOYC) is an evidence-based, eight-session life skills curriculum designed to reduce risk-taking behaviors related to HIV/STI transmission and teen pregnancy. Woven throughout FOYC is a decision-making model that provides guidance and practice in problem solving with a focus on how to obtain factual information on sexual health.
  CImPACT is a single-session intervention including a 24-min educational video filmed in The Bahamas. The video focuses on effective parent-adolescent communication and listening strategies related to difficult topics including "safe-sex" followed by two role-plays for the parent and youth, a discussion, and a condom demonstration.

SUMMARY:
This is a five-year hybrid type 3 effectiveness-implementation study evaluating multilevel strategies to sustain a nationwide implementation of an evidence-based HIV prevention curriculum in schools. Advanced machine learning methods are being used to enhance implementation strategies. A Sequential, Multiple Assignment, Randomized Trial (SMART) design will be employed.

DETAILED DESCRIPTION:
A hybrid type 3 effectiveness-implementation study is proposed, using a SMART adaptive implementation trial that will evaluate the value of multilevel strategies to sustain Focus on Youth in Caribbean + Caribbean Informed Parents and Children Together (FOYC+CImPACT) in schools and harness advanced machine learning to help promote the FOYC+CImPACT sustainability by iteratively enriching implementation strategies. This study will also identify the most effective implementation strategy for teachers who implement <80% of core activities and for adolescents who are unlikely to respond to FOYC+CImPACT by using machine learning approaches. The primary outcome is program sustainability. Data from teachers, students, and focus groups will provide information on inner and outer contexts, strategies to promote implementation and sustainability, and program effectiveness.

Primary implementation of FOYC+CImPACT will be conducted by 156 grade-6 teachers in 65 government primary schools across four years. Annual FOYC booster sessions for students will be conducted by 49 Health and Family Life Education (HFLE) teachers in 30 junior high schools. Approximately 3,500 students will complete the full curricular assessment survey at the beginning and end of grade 6 and at the end of grades 7, 8, and 9.

ELIGIBILITY:
Inclusion Criteria:

* Grade 6 teachers who teach Health and Family Life Education (HFLE) and their classes in 65 government primary schools.
* Grade 7-9 HFLE teachers and their classes in 30 middle schools across 12 Bahamian islands.
* FOYC (Focus on Youth in the Caribbean) is delivered as part of the standard HFLE curriculum.
* Students who: 1) are enrolled in one of the participating schools as general education students in grade 6 (and followed through grades 7-9); and 2) speak and read English.

Exclusion Criteria:

* Students who chose to opt out of participating in the study
* Students who do not speak or read English sufficiently to participate in study activities.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3705 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Fidelity of Implementation | Years 1, 2, 3, and 4
  Adherence to the core activities (number of core activities taught as intended)
Sustainability | Year 4
  Teachers' continued implementation of the intervention with fidelity (at least 80% of core activities) and adherence to program principles across 4 years
Sustainment determinants | Years 1 and 3
  The Sustainment Measurement System Scale (SMSS) is a 35-item instrument that evaluates sustainment determinants and outcomes (one sustainment outcome subscale and seven determinant domain subscales).
  Items are rated on a 5-point scale, from 1 = Little or no extent to 5 = Great extent.
  Subscale scores are calculated as the average of the items within the subscale, ranging from 1 to 5. Higher scores on all subscales indicate greater agreement with the subscale.
Inner and outer context factors affecting implementation | Yeasr 1 and 3
  The Program Sustainability Assessment Tools (PSAT) is an eight-domain, 40-item instrument that assesses a program's capacity for sustainability.
  Items are rated on a 7-point scale from 1 = Little or no extent to 7 = A very great extent.
  Scores are first averaged within each domain, and an overall sustainability score is calculated by averaging the domain scores (range: 1-7). Higher scores indicate a great level of sustainability capacity.
School implementation climate | Years 1 and 3
  The School Implementation Climate Scale (SICS) is a seven-domain, 21-item instrument assessing a school's climate for implementing an evidence-based practice.
  Items are rated on a 5-point scale (0 = Not at all; 4 = Very great extent). Scores are first averaged within each domain, and an overall sustainability score is calculated by averaging the domain scores (range: 0-4). Higher scores indicate a more favorable implementation climate.
Condom use skills | Years 1, 2, 3, and 4
  The Condom-Use Skills Checklist is an 8-item scale assessing youth's understanding of correct condom use.
  Each item is answered True/False. Scores are calculated as the total number of correct responses. Scores range from 0 to 8, with higher scores indicating greater knowledge of condom-use skills.
Self-efficacy | Years 1, 2, 3, and 4
  A 5-item self-efficacy for condom use scale will be utilized to assess students' self-perceived ability to use condoms.
  Items are rated on a 5-point scale (1 = Strongly disagree; 5 = Strongly agree). Scores are calculated as the average of all items, with a range of 1 to 5. Higher scores indicate greater self-efficacy for condom use.
Condom use | Years 1, 2, 3, and 4
  Self-reported condom use in the last sexual intercourse and frequency of condom use in general (always, often, sometimes, or never)

SECONDARY OUTCOMES:
Youth risk and protective behaviors | Years 1, 2, and 4
  The Health-Risk and Protective Factors (HRPF) survey
Youth sensation seeking | Years 1, 2, 3, and 4
  The Health-Risk and Protective Factors (HRPF) survey
Neighborhood risk | Years 1, 2, 3, and 4
  The Health-Risk and Protective Factors (HRPF) survey

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- HIV/AIDS Office, FOY program, Nassau, The Bahamas

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data